CLINICAL TRIAL: NCT05446129
Title: A Phase I Open Label Study to Assess Safety, Feasibility, Efficacy, and Biological Activity of Single Administration of Neoadjuvant Treatments Ezabenlimab in Combination With BI 765063 and Pembrolizumab in Combination With BI 765063 in Patients With Newly Diagnosed Surgically-resectable, Locoregional Colorectal Cancer
Brief Title: A Study in People With Colorectal Cancer to Test Whether Ezabenlimab or Pembrolizumab in Combination With BI 765063 Lead to Side Effects or Delays in Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1502-0001
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Ezabenlimab + BI 765063 (Experimental)
  Interventions: Drug: Ezabenlimab; Drug: BI 765063
- Cohort B: Pembrolizumab + BI 765063 (Experimental)
  Interventions: Drug: BI 765063; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Ezabenlimab — Ezabenlimab
  Arms: Cohort A: Ezabenlimab + BI 765063
Drug: BI 765063 — BI 765063
Drug: Pembrolizumab — Pembrolizumab
  Arms: Cohort B: Pembrolizumab + BI 765063

SUMMARY:
This study is open to people with newly diagnosed colorectal cancer. People who are scheduled for surgery can participate. People either get a medicine called BI 765063 combined with ezabenlimab or combined with pembrolizumab in preparation of the upcoming surgery. The tested medicines in this study are antibodies that may help the immune system fight cancer.

The purpose of this study is to find out how well people with early colorectal cancer can tolerate treatment with these medicines. The study also looks at whether the tumor changes.

Participants are put into 2 groups. One group gets ezabenlimab and BI 765063. The other group gets pembrolizumab and BI 765063. All participants receive the study medicines as 2 subsequent infusions into a vein on a single day.

Participants are in the study for about 4 months. During this time, they visit the study site about 5 times. The doctors check the health of the participants and note any health problems that could have been caused by ezabenlimab, pembrolizumab, or BI 765063. The doctors also check whether these health problems lead to a delay of the planned surgery.

ELIGIBILITY:
Inclusion criteria

* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial. Ability to understand and the willingness to sign a written informed consent.
* Male or female aged = 18 years at the time of informed consent form (ICF) signature.
* Patients with histological diagnosis of resectable colorectal Cancer (CRC), or radiographic/visual findings highly suggestive, with planned confirmatory biopsy.
* CRC lesions must be at least 1 centimeter (cm) in largest diameter and amenable to endoscopic biopsy.
* Patient must be willing and able to have endoscopic biopsy (Goal 3-6 core-needle or surgical/endoscopic biopsies, final number to be determined by the physician performing the procedure as safe) of tumor prior to initiation of therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1. The exception will be patients with long term disability (such as cerebral palsy) that is unlikely to significantly affect their response to therapy.
* Patient is determined to be a surgical candidate for resection of their tumor.
* Adequate organ and marrow function as defined in the protocol.
* Further inclusion criteria apply.

Exclusion criteria

* Patients who are deemed to be at high risk for colonic obstruction and/or perforation per investigator assessment.
* Patients eligible for neoadjuvant therapy (chemotherapy, radiotherapy, chemoradiotherapy) as standard of care.
* Major surgery (major according to the investigator's assessment) performed within 4 weeks prior to administration of trial medication.
* Patients who must or wish to continue the intake of restricted medications (as defined in the protocol) or any drug considered likely to interfere with the safe conduct of the trial.
* Patients not expected to comply with the protocol requirements or not expected to complete the trial as scheduled (e.g. chronic alcohol or drug abuse or any other condition that, in the investigator's opinion, makes the patient an unreliable trial participant).
* Previous enrolment in this trial.
* Currently enrolled in another investigational device or drug trial, or less than 30 days since ending another investigational device or drug trial(s) or receiving other investigational treatment(s).
* Patients who have had chemotherapy or radiotherapy within 6 months prior to entering the study for a different primary tumor, or those that have received locoregional therapy (radiation, chemoembolization, etc.) for the target lesion that will be biopsied and subsequently resected. Previous therapy for a different cancer (a different primary) is acceptable.
* Prior immune checkpoint inhibitor therapy.
* Patients with metastatic or recurrent disease, for which the intent of surgery would not be curative.
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https:// www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label, single-center, two-arm, parallel-group Phase I trial to assess the safety and feasibility of a single dose of BI 765063 in combination with either ezabenlimab (Cohort A) or pembrolizumab (Cohort B) in participants with early-stage, resectable colorectal cancer in a neoadjuvant setting.
Pre-assignment Details: Only two participants were enrolled in this trial. All participants were screened for eligibility prior to participation and attended a specialist site to ensure strict adherence to all inclusion criteria and none of the exclusion criteria. Participants were not allocated to a treatment group if any entry criteria were violated. The trial was prematurely discontinued due to the low number of enrolled participants.
Groups:
- Cohort A: Ezabenlimab + BI 765063: Participants received two separate consecutive intravenous (i.v.) infusions on Day 1. First, they received one flat dose of 240 milligram (mg) ezabenlimab and then one dose of BI 765063.
- Cohort B: Pembrolizumab + BI 765063: Participants received two separate consecutive intravenous (i.v.) infusions on Day 1. First, they received one flat dose of 200 milligram (mg) Pembrolizumab and then one dose of BI 765063.
Period: Overall Study
Arm/Group | Cohort A: Ezabenlimab + BI 765063 | Cohort B: Pembrolizumab + BI 765063
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: As only two participants were enrolled in the study, analysis sets were not defined.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Ezabenlimab + BI 765063 | Cohort B: Pembrolizumab + BI 765063 | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Customized [Count of Participants; unit: Participants]
  >= 18 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint: Proportion of Patients With at Least One Occurrence of a Safety or Feasibility Event
Description: Safety:
  A safety event was defined as any grade 3 or higher adverse events (AEs; according to National Cancer Institute's Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) related to study treatments at any point within the follow-up period following the administration of study treatments.
  Feasibility (delay in surgery):
  A feasibility event or delay in surgery was defined as any treatment related AE leading to delay in surgery, which was scheduled to take place between 2 weeks and up to 6 weeks following the study treatment administration will be considered as a relevant AE for this endpoint.
Time Frame: Up to 91 days after drug administration.
Population: The trial was discontinued early due to slow participant enrollment. Only a patient profile listing containing data collected for individual participants was compiled and statistical outputs and analyses i.e. the primary and secondary outcome measurements were not assessed.
Measure: Number; unit: Percentage of Participants
Groups:
- Ezabenlimab + BI 765063: Participants assigned to this Cohort received a flat dose of 240 mg ezabenlimab in combination with a dose of BI 765063.
- Pembrolizumab + BI 765063: Participants assigned to this Cohort received a flat dose of 200 mg pembrolizumab in combination with a dose of BI 765063.
Arm/Group | Ezabenlimab + BI 765063 | Pembrolizumab + BI 765063
Number analyzed (Participants) | 1 | 1
Percentage of Participants | 0 | 0

2. Secondary Outcome: Pathologic Response (PR)
Description: At least 50% or more tumor regression classified as per Mandard tumor regression grading system, in viable adenocarcinoma cells in the surgical specimen, including lymph nodes. Pathological response includes complete pathology response (CR), near complete pathological response (near CR) and partial pathological response
Time Frame: Up to 91 days after drug administration.
Population: The trial was discontinued early due to slow participant enrollment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ezabenlimab + BI 765063 | Pembrolizumab + BI 765063
Number analyzed (Participants) | 1 | 1
Percentage of Participants
  Complete pathology response (CR) | 0 | 0
  Near complete pathological response (near CR) | 0 | 0
  Partial pathological response | 0 | 0
  No response | 1 [NA to NA] — Not calculable with one subject | 1 [NA to NA] — Not calculable with one subject

3. Secondary Outcome: Time From Administration of Trial Treatment to Surgery
Description: Time from administration of trial treatment to surgery, defined as the time in days that elapses between administration of neoadjuvant trial therapy and surgical resection.
Time Frame: Up to 91 days after drug administration.
Population: The trial was discontinued early due to slow participant enrollment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ezabenlimab + BI 765063 | Pembrolizumab + BI 765063
Number analyzed (Participants) | 1 | 1
days | 19 (NA) — The standard deviation for this endpoint could not be calculated. | 19 (NA) — The standard deviation for this endpoint could not be calculated.

4. Secondary Outcome: Radiographic Response Rate
Description: Radiographic response on pre-surgical imaging, following receipt of the neoadjuvant therapy, as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). The same imaging procedure(s) (computed tomography, magnetic resonance imaging scan) were used throughout the trial.
Time Frame: Up to 91 days after drug administration.
Population: The trial was discontinued early due to slow participant enrollment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ezabenlimab + BI 765063 | Pembrolizumab + BI 765063
Number analyzed (Participants) | 1 | 1
Percentage of participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 0 | 0
  Progressive Disease (PD) | 0 | 0
  Stable Disease (SD) | 100 [NA to NA] — Not calculable with one subject | 100 [NA to NA] — Not calculable with one subject

ADVERSE EVENTS:
Time Frame: Up to 91 days after drug administration.
Description: All participants that had been screened and treated, and had completed the trial before the trial was discontinued.
Arm/Group | Ezabenlimab + BI 765063 | Pembrolizumab + BI 765063
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ezabenlimab + BI 765063 (N=1) | Pembrolizumab + BI 765063 (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The trial was terminated early due to the sponsor's decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT05446129/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT05446129/SAP_001.pdf